CLINICAL TRIAL: NCT06795451
Title: Modulating Spinal Interoceptive Pathways to Evaluate Their Role and Therapeutic Potential in MDD Symptomatic Domains
Acronym: MOSPID
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Francisco Romo-Nava, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0510; 1R61MH133770-01A1 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Depression - Major Depressive Disorder
Keywords: depression; non-invasive; neuromodulation; spinal stimulation; transcutaneous spinal direct current stimulation; major depressive disorder; interoception; spinal interoceptive pathways; laser-evoked potentials
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- 2.0 Sham (Sham Comparator): Sham will also be compared to "No intervention"
  Interventions: Device: transcutaneous spinal direct current stimulation
- 2.5 Active (Active Comparator)
  Interventions: Device: transcutaneous spinal direct current stimulation
- 3.0 Active (Active Comparator)
  Interventions: Device: transcutaneous spinal direct current stimulation
- 3.5 Active (Active Comparator)
  Interventions: Device: transcutaneous spinal direct current stimulation

INTERVENTIONS:
Device: transcutaneous spinal direct current stimulation — transcutaneous spinal direct current stimulation

SUMMARY:
Spinal interoceptive pathways (SIPs) convey bodily signals to an interoceptive system in the brain and their dysregulation is linked to major depressive disorder (MDD). Current treatments are partially effective and the role of SIPs in MDD is vastly unexplored. Preliminary data suggests that SIPs are feasible therapeutic targets in MDD. The central hypothesis is that non-invasive spinal cord stimulation will modulate SIPs to elucidate their role and therapeutic potential in MDD using an R61/33 phased innovation approach.

R61 phase specific aims (SA). The specific goal will be to evaluate spinal and brain-based SIPs target engagement markers of transcutaneous spinal direct current stimulation (tsDCS) in MDD with two SAs: SA1) To determine tsDCS SIPs modulation using laser-evoked potentials (LEPs) as electroencephalography (EEG)- based neural measures of target engagement. SA2) To evaluate optimal tsDCS dose based upon tolerability and SIPs target engagement markers. Anodal tsDCS will be evaluated as a tool to modulate SIPs in MDD. SIPs (Aδ and C fibers) can be evaluated via LEPs as neural measures (EEG) elicited in MDD-relevant brain regions within an interoceptive system. Prior data shows anodal tsDCS inhibits SIPs and LEPs N2 component will be assessed as tsDCS engagement markers. Adults with MDD (n=67) will participate in a double-blind, crossover, sham-controlled study to evaluate tsDCS at 0,2.5,3, and 3.5 mA. The working hypothesis is that tsDCS will induce a change in LEPs (SA1) in a dose-dependent and tolerable manner (SA2), supporting their use as SIPs engagement markers. Go/No-Go milestones: Compared to sham, the active tsDCS dose that induces a change in LEPs at a preestablished threshold will be evidence of SIPs engagement and "Go" criteria for the R33 phase.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 yrs., inclusive,
* Female or Male,
* With current MDD episode according to MINI 7.0.2. duration (≥4 weeks and

  ≤ 2 yrs.),
* Current BMI ≥18.5 and ≤ 35 kg/mts2, inclusive,
* MADRS score at screening ≥18
* Currently on an FDA- approved antidepressant medication at a stable therapeutic dose for ≥ 8 weeks,
* Psychotherapeutic interventions are allowed if dose/frequency stable for ≥4 weeks,
* Anxiety disorders allowed if no more than moderate in severity and are not the main diagnosis,
* Using an effective contraceptive method (participants with childbearing potential), and 10)Able to complete study related tasks.

Exclusion Criteria:

* Treatment resistance during current depressive episode (>2 treatment trials at adequate doses/duration), including medication and neuromodulation treatments.
* Current/lifetime diagnosis of bipolar disorder or schizophrenia spectrum disorders.
* Significant risk of suicide according to CSSRS or clinical judgment, or suicidal behavior in the past year.
* Psychotic symptoms during the current MDD episode or in the past 6 months.
* Current (past month) substance use disorder (nicotine, caffeine allowed).
* Current unstable neurological conditions including seizure disorders (infantile seizures are not exclusionary), neurodegenerative disorders, or stroke.
* Evidence of severe peripheral neuropathy.
* History of moderate to severe traumatic brain injury (e.g., skull fracture or loss of consciousness >10 minutes) or spinal cord injury.
* Unstable clinically significant medical conditions (e.g., uncontrolled hypertension as indicated by a systolic >150 mmHg or diastolic >95mmHg).
* History of cancer allowed if remitted for the past 5 years.
* Use of anticonvulsant medications and calcium channel blockers at screening.
* Current severe pain conditions or need for chronic use of pain medication including NSAIDs and opiates.
* Implanted electronic medical devices.
* Neuromodulation interventions in the past month.
* Active skin lesions on electrode placement sites.
* pregnant or breastfeeding.
* Suspected IQ <80.
* Any other relevant clinical reason as judged by the clinician.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
N2 peak amplitude | 5 weeks
  Peak amplitude change in N2 expressed in sham to active percentage of change.
N2 latency | 5 weeks
  The N2 latency sham to active tsDCS time change in milliseconds (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Romo-Nava, MD, PhD, Principal Investigator — Lindner Center of Hope/ University of Cincinnati
Locations (1):
- Lindner Center of Hope, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to NIMH Data sharing plan and uploaded to a data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of primary statistical plan and unblinding of data.
Access Criteria: Deidentified data will be shared on a biorepository.

REFERENCES:
- [Background] Romo-Nava F, Awosika OO, Basu I, Blom TJ, Welge J, Datta A, Guillen A, Guerdjikova AI, Fleck DE, Georgiev G, Mori N, Patino LR, DelBello MP, McNamara RK, Buijs RM, Frye MA, McElroy SL. Effect of non-invasive spinal cord stimulation in unmedicated adults with major depressive disorder: a pilot randomized controlled trial and induced current flow pattern. Mol Psychiatry. 2024 Mar;29(3):580-589. doi: 10.1038/s41380-023-02349-9. Epub 2023 Dec 20. PMID 38123726